CLINICAL TRIAL: NCT00003729
Title: Phase II Study of Fludarabine + Idarubicin + Aracytine in Refractory or Relapsed ALL in Children
Brief Title: Combination Chemotherapy in Treating Children With Relapsed or Refractory Acute Lymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-58953; EORTC-58953
Record Dates: First submitted 1999-11-01; First posted 2003-12-10 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; L1 childhood acute lymphoblastic leukemia; L2 childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cytarabine; fludarabine phosphate; Idarubicin

INTERVENTIONS:
Drug: cytarabine
Drug: fludarabine phosphate
Drug: idarubicin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating children who have relapsed or refractory acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the complete response rate to combination fludarabine, idarubicin, and cytarabine in children with relapsed or refractory acute lymphocytic leukemia. II. Evaluate the safety and tolerance of this treatment in these patients. III. Evaluate the time to progression, disease free survival, and overall survival of these patients.

OUTLINE: This is an open label, multicenter study. Patients receive idarubicin IV over 1 hour on days 1-3. Fludarabine IV is administered over 30 minutes on days 1-5. Cytarabine IV is administered over 4 hours on days 1-5. If partial response is obtained, patients receive a second course of treatment. Patients receive a consolidation course in the absence of disease progression and unacceptable toxicity. Idarubicin IV is administered over 1 hour on days 1 and 2. Fludarabine IV is administered over 30 minutes, followed by cytarabine IV over 4 hours on days 1-5. Patients are followed every 3 months for 2 years or until death.

PROJECTED ACCRUAL: A total of 24-45 patients will be accrued for this study within 27 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Cytologically diagnosed relapsed or refractory acute lymphocytic leukemia previously treated with front line therapy FAB L1 or L2 Bone marrow relapse either isolated or associated with CNS or testicular relapse Bone marrow blast cells greater than 10% No isolated CNS relapse

PATIENT CHARACTERISTICS: Age: Under 18 Performance status: WHO 0-2 Play-performance scale at least 60% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin less than 2.5 times normal Renal: Creatinine less than 2.5 times normal Cardiovascular: No symptoms of cardiac failure No decline of ejection fraction by more than 20% of the lower limit of normal Shortening fraction at least 25% Other: No psychological, familial, sociological or geographical condition that would hamper compliance No uncontrolled infection

PRIOR CONCURRENT THERAPY: At least 6 months since prior autologous bone marrow transplantation No prior allogeneic bone marrow transplantation No concurrent treatment with other experimental drug

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 1998-12; Primary Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Thyss, MD, Study Chair — Centre Antoine Lacassagne
Locations (23):
- Belgium (7):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - Hopital Universitaire Des Enfants Reine Fabiola, Brussels (Bruxelles)
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels (Bruxelles)
  - Universitair Ziekenhuis Gent, Ghent (Gent)
  - U.Z. Gasthuisberg, Leuven
  - Centre Hospitalier Regional de la Citadelle, Liege (Luik)
  - Clinique de l'Esperance, Montegnée
- France (15):
  - Centre Hospitalier Regional et Universitaire d'Angers, Angers
  - CHR de Besancon - Hopital Saint-Jacques, Besançon
  - CHU de Caen, Caen
  - CHR de Grenoble - La Tronche, Grenoble
  - Centre Hospitalier Regional de Lille, Lille
  - Hopital Debrousse, Lyon
  - Hopital Arnaud de Villeneuve, Montpellier
  - CHR Hotel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hopital Robert Debre, Paris
  - Institut Curie - Section Medicale, Paris
  - Hopital Jean Bernard, Poitiers
  - Hopital Americain, Reims
  - Hopital Universitaire Hautepierre, Strasbourg
  - Hopital des Enfants (Purpan Enfants), Toulouse
- Hospital Escolar San Joao, Porto, Portugal